CLINICAL TRIAL: NCT05619536
Title: A Phase 1, Randomized, Double-Blind, Single Ascending Dose Study to Determine the Safety, Tolerability, and Pharmacokinetics of CD388 Subcutaneous Administration in Healthy Japanese Subjects
Brief Title: Study of CD388 Subcutaneous Administration in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD388.SQ.1.03
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 9 subjects randomized in a 7:2 ratio to receive either 50 mg CD388 SQ injection or matching placebo injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 2 (Experimental): 9 subjects randomized in a 7:2 ratio to receive either 150 mg CD388 SQ injection or matching placebo injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo
- Cohort 3 (Experimental): 9 subjects randomized in a 7:2 ratio to receive either 450 mg CD388 SQ injection or matching placebo injection
  Interventions: Combination Product: CD388 Injection; Drug: Saline placebo

INTERVENTIONS:
Combination Product: CD388 Injection — CD388 liquid for injection
Drug: Saline placebo — Sterile normal saline for injection

SUMMARY:
The purpose of this study is to determine the safety and tolerability profile of CD388 Injection, as compared to saline placebo, when dosed by subcutaneous (SQ) administration as a single dose to healthy Japanese adult subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, prospective, randomized, double-blind study of ascending single doses of CD388 Injection administered SQ to healthy Japanese adult subjects. The goals are to assess safety, tolerability, and pharmacokinetics (PK) of CD388.

ELIGIBILITY:
Inclusion Criteria:

1. Must be of Japanese descent with Japanese parents and grandparents, as determined by subject's verbal report.
2. Willing and able to provide written informed consent.
3. Males and females 18 to 65 years of age, inclusive.
4. A female subject must meet one of the following criteria:

   1. If of childbearing potential - agrees to use a highly effective, preferably user-independent method of contraception (failure rate of <1 percent per year when used consistently and correctly) for at least 30 days prior to screening and agrees to remain on a highly effective method until 7 months after last dose of study medication, whichever is longer. Examples of highly-effective methods of contraception include: abstinence from heterosexual intercourse; hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch); intrauterine device (with or without hormones); or a double barrier method (e.g., condom and spermicide).
   2. If a female of non-childbearing potential - should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion without reversal surgery) or in a menopausal state (at least 1 year without menses), as confirmed by follicle-stimulating hormone (FSH) levels (≥40 milli-International units [mIU]/milliliter [mL]).
5. A woman of childbearing potential must have a negative highly sensitive serum pregnancy test (β-human chorionic gonadotropin) at screening and a negative urine pregnancy test on Day -1 before the first dose of study drug.
6. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of at least 7 months after study drug administration.
7. A male subject that engages in sexual activity that has the risk of pregnancy must agree to use a double barrier method (e.g., condom and spermicide) and agree to not donate sperm during the study and for at least 7 months after the last dose of the study medication.
8. Good health and without signs or symptoms of current illness.
9. Normal clinical examination, including:

   1. No physical examination findings that an Investigator determines would interfere with interpretation of study results.
   2. Screening ECG without clinically significant abnormalities.
   3. Creatinine clearance (CrCL) ≥80 mL/minute as calculated using the Cockcroft-Gault equation.
   4. Negative urine screen for drugs of abuse and alcohol at screening and Day -1.
10. Body weight ≥50 kilograms (kg) and body mass index (BMI; calculated as weight in kg divided by height in meters [m] squared) between 18.0 and 30.0 kg/m^2, inclusive.
11. Willing to refrain from strenuous physical activity that could cause muscle aches or injury, including contact sports, at any time from screening through 30 days after any dose of study drug.
12. Subject has adequate venous access for blood collection.

Exclusion Criteria:

1. History of any hypersensitivity or allergic reaction to zanamivir or other neuraminidase inhibitors (i.e., laninamivir, oseltamivir, peramivir), or to excipients of the CD388 Injection drug formulation; or history of drug-induced exfoliative skin disorders (e.g., Stevens-Johnson syndrome [SJS], erythema multiforme, or toxic epidermal necrolysis [TEN]).
2. History of any of the following:

   1. Allergies, anaphylaxis, skin rashes (foods such as milk, eggs, medications, vaccines, polyethylene glycol [PEG], etc.).
   2. Chronic immune-mediated disease, positive first-degree family history of autoimmune diseases.
   3. Atopic dermatitis or psoriasis.
   4. Bleeding disorder.
   5. Psychiatric condition, seizures, hallucinations, anxiety, depression, or treatment for mental conditions.
   6. Migraines.
   7. Syncope, or vasovagal syndrome with injections or blood draws.
   8. Cardiac arrhythmia considered clinically significant by the Investigator.
3. Subjects with one or more of the following laboratory abnormalities at screening as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events v2.1 (DAIDS 2017):

   1. Serum creatinine, Grade ≥1 (≥1.1 × upper limit of normal [ULN]).
   2. Pancreatic amylase or lipase, Grade ≥2 (≥1.5 × ULN).
   3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT), Grade ≥1 (≥1.25 × ULN).
   4. Total bilirubin, Grade ≥1 (≥1.1 × ULN).
   5. Any other toxicity Grade ≥2, except for Grade 2 elevations of triglycerides, low density lipoprotein cholesterol, and/or total cholesterol.
   6. Any other laboratory abnormality considered to be clinically significant by the Investigator.

      * Note: Retesting of abnormal laboratory values that may lead to exclusion will be allowed once without prior asking approval from the Sponsor. Retesting will take place during a scheduled or unscheduled visit during screening. Subjects with a normal value at retest may be included.
4. Alcohol or drug addiction in the past 2 years.
5. Experiencing symptoms of acute illness or chronic disease within 14 days prior to clinical research unit (CRU) check-in.
6. At screening, a positive result for hepatitis B virus surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody.
7. A positive result at CRU check-in for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by polymerase chain reaction (PCR).
8. Unwilling to comply with local health policy effective at the time regarding coronavirus disease 2019 (COVID-19). Full COVID-19 vaccination prior to participation is strongly recommended.
9. Women who are pregnant or nursing.
10. Received any over-the-counter (OTC) medications or nutritional supplements within 7 days, or any prescription medications within 14 days or <5 half-lives prior to dosing, whichever is longest (except for hormonal contraceptives, acetaminophen, or ibuprofen).
11. Current nicotine user or has quit habitual nicotine use in the 30 days prior to screening.
12. Received any vaccines or immunoglobulins within 28 days prior to dosing (90 days in case of intravenous immunoglobulin [IVIg] or biologics, or 14 days for COVID-19 vaccine).
13. Donated blood (within 56 days of screening) or plasma (within 7 days of screening) or experienced significant blood loss or significant blood draw (blood donation or blood loss ≥500 mL) when participating in non-interventional clinical trials within 30 days prior to dosing.
14. Received a blood transfusion within 28 days prior to dosing.
15. Received any biologics within 90 days prior to dosing; or previous participation in another study (including investigational device studies) within 30 days of dosing or 5 half-lives of the study drug, whichever is longer, prior to screening (prior participation at any time in non-invasive methodology trials in which no drugs were given is acceptable).
16. Previous treatment with CD388.
17. Preplanned surgery at any time during the study.
18. The Principal Investigator (PI) considers that the volunteer should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Equils, MD, Study Director — Cidara Therapeutics Inc.; Youngjun Kim, MD, Principal Investigator — Altasciences Clinical Los Angeles, Inc.
Locations (1):
- Altasciences Clinical Los Angeles, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned total enrollment was 27 participants. One participant in the 150 milligram (mg) CD388 arm withdrew consent shortly after dosing and was replaced, resulting in an overall enrollment of 28 participants.
Groups:
- 50 mg CD388: 7 participants randomized to receive a single dose of 50 mg CD388 via subcutaneous (SQ) injection
  CD388 Injection: CD388 liquid for injection
- 150 mg CD388: 8 participants randomized to receive a single dose of 150 mg CD388 via SQ injection
  CD388 Injection: CD388 liquid for injection
- 450 mg CD388: 7 participants randomized to receive a single dose of 450 mg CD388 via SQ injection
  CD388 Injection: CD388 liquid for injection
- Pooled Placebo: 6 participants randomized to receive a single dose of saline placebo via SQ injection
  Saline placebo: Sterile normal saline for injection
Period: Overall Study
Arm/Group | 50 mg CD388 | 150 mg CD388 | 450 mg CD388 | Pooled Placebo
Started | 7 | 8 (One participant withdrew consent shortly after dosing with 150 mg CD388 and was replaced; this participant's samples were not analyzed and were not used for the pharmacokinetic (PK) analyses.) | 7 | 6
Completed | 7 | 6 | 6 | 5
Not Completed | 0 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population analyzed consisted of all participants who received any amount of study drug.
Groups:
- 50 mg CD388: 7 participants randomized to receive a single dose of 50 mg CD388 via SQ injection
  CD388 Injection: CD388 liquid for injection
- Total: Total of all reporting groups
Arm/Group | 50 mg CD388 | 150 mg CD388 | 450 mg CD388 | Pooled Placebo | Total
Number analyzed (Participants) | 7 | 8 | 7 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (13.60) | 50.4 (11.90) | 46.0 (15.35) | 49.8 (15.99) | 49.4 (13.49)
Age, Continuous [Median (Full Range); unit: years] | 54.0 [22 to 62] | 55.0 [26 to 64] | 47.0 [21 to 65] | 54.5 [20 to 63] | 54.0 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 2 | 12
  Male | 2 | 5 | 5 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 7 | 6 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 8 | 7 | 6 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 7 | 6 | 28
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 62.84 (7.917) | 69.71 (11.421) | 73.27 (14.517) | 68.55 (7.073) | 68.64 (10.884)
Weight [Median (Full Range); unit: kg] | 61.50 [52.5 to 74.9] | 74.10 [51.8 to 84.9] | 77.10 [51.7 to 90.9] | 66.10 [61.1 to 77.6] | 67.15 [51.7 to 90.9]
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 163.71 (7.607) | 166.03 (6.489) | 170.57 (8.646) | 170.97 (8.400) | 167.64 (7.931)
Height [Median (Full Range); unit: cm] | 161.20 [155.1 to 174.5] | 166.70 [156.0 to 173.2] | 173.30 [157.6 to 178.3] | 173.25 [156.0 to 179.7] | 169.20 [155.1 to 179.7]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/meter^2 (kg/m^2)] | 23.46 (2.938) | 25.20 (3.400) | 24.94 (3.009) | 23.57 (3.153) | 24.35 (3.068)
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 22.70 [20.2 to 29.4] | 25.50 [20.3 to 30.0] | 24.80 [20.4 to 28.6] | 23.90 [19.7 to 27.4] | 24.25 [19.7 to 30.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs) After a Single Dose of CD388
Description: Number of TEAEs reported, including but not limited to adverse events (AEs) and serious adverse events (SAEs) (including systemic reactogenicity/injection site reactions and hypersensitivity reactions), and AEs leading to study drug discontinuation and/or study withdrawal, based on vital signs, electrocardiogram (ECG), and clinical laboratory test (including hematology, coagulation, serum chemistry, and urinalysis) abnormalities following a single dose of CD388.
Time Frame: From Day 1 through the final study visit (Day 120 for the 50 mg dose arm; Day 165 for all others)
Population: The Safety Population included all participants who received any amount of study drug.
Measure: Number; unit: events
Arm/Group | 50 mg CD388 | 150 mg CD388 | 450 mg CD388 | Pooled Placebo
Number analyzed (Participants) | 7 | 8 | 7 | 6
events | 7 | 3 | 6 | 2

2. Primary Outcome: Severity of Treatment-Emergent Adverse Events (TEAEs) After a Single Dose of CD388
Description: Severity of TEAEs reported, including but not limited to adverse events (AEs) and serious adverse events (SAEs) (including systemic reactogenicity/injection site reactions and hypersensitivity reactions), and AEs leading to study drug discontinuation and/or study withdrawal, based on vital signs, electrocardiogram (ECG), and clinical laboratory test (including hematology, coagulation, serum chemistry, and urinalysis) abnormalities following a single dose of CD388.
Time Frame: From Day 1 through the final study visit (Day 120 for the 50 mg dose arm; Day 165 for all others)
Population: The Safety Population included all participants who received any amount of study drug.
Measure: Number; unit: events
Arm/Group | 50 mg CD388 | 150 mg CD388 | 450 mg CD388 | Pooled Placebo
Number analyzed (Participants) | 7 | 8 | 7 | 6
events
  Grade 1 (Mild) | 7 | 3 | 6 | 2
  Grade 2 (Moderate) | 0 | 0 | 0 | 0
  Grade 3 (Severe) | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) Following CD388 Injection Administration
Description: Evaluation of the maximum plasma concentration (Cmax) following subcutaneous administration of a single dose of CD388.
Time Frame: At inpatient visits on Days 1, 2, 3, 4, 5, 6, 7, 9, 11, and 14; and at outpatient visits on Day 30 (±3 days), Day 45 (±3 days), Day 60 (±5 days), Day 90 (±7 days), and either Day 120 (±14 days) (Cohort 1 only) or Day 165 (±14 days) (Cohorts 2 and 3 only)
Population: The Pharmacokinetic (PK) Analysis Population included all participants who received a CD388 injection with at least one post-dose time point sampling. Participants who did not complete the sampling schedule may be included in the PK analysis for only the PK parameters that were judged not to be affected by the missing sample(s).
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (ug/mL)
Groups:
- Cohort 1: Participants randomized to receive a single SQ injection of 50 mg CD388
- Cohort 2: Participants randomized to receive a single SQ injection of 150 mg CD388
- Cohort 3: Participants randomized to receive a single SQ injection of 450 mg CD388
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
micrograms/milliliter (ug/mL) | 3.87 (0.776) | 13.5 (4.10) | 41.7 (9.27)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) Following CD388 Injection Administration
Description: Evaluation of the time to maximum plasma concentration (Tmax) following subcutaneous administration of a single dose of CD388.
Time Frame: as for outcome 3
Population: The PK Analysis Population included all participants who received a CD388 injection with at least one post-dose time point sampling. Participants who did not complete the sampling schedule may be included in the PK analysis for only the PK parameters that were judged not to be affected by the missing sample(s).
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
hours (h) | 312.00 [192.00 to 313.03] | 97.00 [48.00 to 313.00] | 144.00 [72.00 to 312.02]

5. Secondary Outcome: Terminal Elimination Half-life (t½) Following CD388 Injection Administration
Description: Evaluation of the terminal elimination half-life (t½) following subcutaneous administration of a single dose of CD388.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
hours (h) | 1325.86 (289.24) | 1284.26 (389.61) | 1210.10 (193.31)

6. Secondary Outcome: Apparent Clearance (CL/F) Following CD388 Injection Administration
Description: Evaluation of the apparent clearance (CL/F) following subcutaneous administration of a single dose of CD388.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
liters/hour (L/h) | 0.00653 (0.000529) | 0.00723 (0.00200) | 0.00764 (0.00144)

7. Secondary Outcome: Apparent Volume of Distribution (VZ/F) Following CD388 Injection Administration
Description: Evaluation of the apparent volume of distribution (VZ/F) following subcutaneous administration of a single dose of CD388.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
liters (L) | 12.5 (2.87) | 12.6 (3.42) | 13.3 (3.10)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Quantifiable Sample (AUC[0-last]) Following CD388 Injection Administration
Description: Evaluation of the area under the plasma concentration-time curve from time 0 to time of last quantifiable sample (AUC[0-last]) following subcutaneous administration of a single dose of CD388.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
ug*h/mL | 5880 (615) | 18900 (5730) | 53300 (8320)

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC[0-∞]) Following CD388 Injection Administration
Description: Evaluation of the area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC[0-∞]) following subcutaneous administration of a single dose of CD388.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 7 | 7
ug*h/mL | 7700 (657) | 22200 (6390) | 60600 (10700)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants from the time of signing the informed consent form through the final study visit (Day 120 for the 50 mg dose arm; Day 165 for all others).
Description: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were assessed in the Safety Population, which included all participants who received any amount of the study drug.
Arm/Group | 50 mg CD388 | 150 mg CD388 | 450 mg CD388 | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 3/8 | 7/7 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg CD388 (N=7) | 150 mg CD388 (N=8) | 450 mg CD388 (N=7) | Pooled Placebo (N=6)
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0
Injection site hemorrhage (General disorders) | 0 | 0 | 2 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT05619536/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT05619536/SAP_001.pdf